CLINICAL TRIAL: NCT02003196
Title: Effects of Viral Reactivation on Outcomes of Brain-injured Patients ( IBIS-VIRUS)
Acronym: IBIS-VIRUS
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC13_0228
Record Dates: First submitted 2013-12-02; First posted 2013-12-06 (Estimated); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Brain Injury
Keywords: Brain injury; virus; immunosuppression; mechanical ventilation
MeSH Terms: conditions — Brain Injuries; Virus Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Morbidity and mortality of ICU patients is increased by the development of a "immunosuppression" systemic (IS). This IS develops in the early hours of hospitalization and is responsible for severe infections, including viral reactivations (Cytomegalovirus or Herpes Simplex Virus). Viral reactivation was associated with increased morbidity and mortality in intensive care units. In clinical practice, they are searched at the onset of organ failure or unexplained fever. The investigators wish to conduct this research in the stroke patients to assess the predictive power of these viral reactivations on the duration of mechanical ventilation.

DETAILED DESCRIPTION:
PCR for herpes simplex virus in blood and in tracheal aspirate (Day-1, Day-7 and Day-15) - clinicians are blinded to the results PCR for Cytomegalovirus in blood and in tracheal aspirate (Day-1, Day-7 and Day-15) - clinicians are blinded to the results

ELIGIBILITY:
Inclusion Criteria:

* Hospitalisation in intensive care unit
* Acute brain injury (trauma, subarachnoid haemorrhage, stroke, infection) with Glasgow Coma Scale <= 12
* Age between 18 and 75 years
* Mechanical ventilation > 24 hours

Exclusion Criteria:

* encephalopathy post anoxy
* active cancer
* Immunosuppresseur treatment
* pregnancy
* history of autoimmune disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Acute brain injury (trauma, subarachnoid haemorrhage, stroke, infection) with Glasgow Coma Scale <= 12
  * Age between 18 and 75 years
Sampling Method: Probability Sample
Enrollment: 375 (Actual)
Dates: Start 2014-01-05 (Actual); Primary Completion 2020-03-26 (Actual); Study Completion 2020-03-26 (Actual)

PRIMARY OUTCOMES:
Ventilatory-free days at day 90 | 90 days

SECONDARY OUTCOMES:
Bacterial hospital acquiered infection | 28 days
organ failure | 28 days
hospitalisation length of stay | 28 days
Mortality | 28 days and 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Karim Asehnoune, Pr, Principal Investigator — Nantes University Hospital
Locations (1):
- CHU de Nantes, Nantes, France

REFERENCES:
- [Derived] Anani H, Destras G, Regue H, Bulteau S, Bressollette-Bodin C, Roquilly A, Josset L. Metagenome-assembled complete genome of Bohxovirus, a virulent bacteriophage involved in the prediction of hospital-acquired pneumonia in intubated critically ill patients. Microbiol Resour Announc. 2025 Dec 11;14(12):e0059225. doi: 10.1128/mra.00592-25. Epub 2025 Oct 29. PMID 41159973
- [Derived] Anani H, Destras G, Bulteau S, Castain L, Semanas Q, Burfin G, Petrier M, Martin FP, Poulain C, Dickson RP, Bressollette-Bodin C, Roquilly A, Josset L. Lung virome convergence precedes hospital-acquired pneumonia in intubated critically ill patients. Cell Rep Med. 2025 Sep 16;6(9):102289. doi: 10.1016/j.xcrm.2025.102289. Epub 2025 Sep 5. PMID 40914165